CLINICAL TRIAL: NCT07280195
Title: ZYNRELEF vs Continuous Catheter for Pain Management Following Shoulder Arthroplasty
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Alexander Aleem, Associate Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202509174
Record Dates: First submitted 2025-11-20; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Total Shoulder Arthroplasty; Pain Management
Keywords: ZYNRELEF; Total shoulder arthroplasty
MeSH Terms: conditions — Agnosia | interventions — bupivacaine-meloxicam drug combination; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ZYNRELEF (Active Comparator)
  Interventions: Drug: Zynrelef
- Interscalene block with continuous catheter pump (Active Comparator)
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Zynrelef — ZYNRELEF
  Arms: ZYNRELEF
Drug: Bupivacaine — Interscalene block with continuous catheter pump
  Arms: Interscalene block with continuous catheter pump

SUMMARY:
The purpose of this study is to determine if local intra-operative application of ZYNRELEF (topical medication) during shoulder replacement surgery improves pain control (as defined by opioid consumption after surgery) compared to the use of an interscalene block with catheter. This is a randomized clinical trial without blinding. Subjects will complete patient reported outcomes before and after surgery. Subjects will track their narcotic use, pain scores and pain satisfaction after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18 years or older
2. Indicated to undergo primary total shoulder arthroplasty (anatomic or reverse)

Exclusion Criteria:

1. Any persons unable to consent, will not be eligible
2. Patients undergoing revision arthroplasty or reverse shoulder arthroplasty
3. Proximal humerus fractures
4. Inability to have interscalene anesthetic catheter placement
5. Compromised baseline renal function (CrCl < 50)
6. BMI > 40
7. History of GI bleed, prior duodenal surgery, or gastric sleeve resection
8. Current narcotic use or prior consistent narcotic exposure in the last 6 months
9. Use of perioperative oral steroid medications
10. Active Workman's compensation claim
11. Prior shoulder arthroplasty on the contralateral side in which an interscalene catheter was used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Narcotic consumption | From surgery to two-weeks following surgery
  Narcotic consumption measured in morphine equivalent units (MEU)

SECONDARY OUTCOMES:
Pain management cost | Perioperative
  Total cost of the interscalene single shot block plus Zynrelef compared to the cost of the block plus catheter with pain pump
Pain management administration | Perioperative
  Time needed by the anesthesiologists to perform the blocks in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Aleem, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No